CLINICAL TRIAL: NCT01735799
Title: THE ASSOCIATION BETWEEN FATTY LIVER (NAFLD) DISEASE AND PCOS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assy Nimer (Other Government)
Responsible Party: Sponsor-Investigator, Assy Nimer, Assy Nimer, Ziv Medical Center, Ziv Hospital
Organization: Ziv Hospital (Other Government)
Other Study IDs: 0068-12-ZIV
Record Dates: First submitted 2012-11-25; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Polycystic Ovarian Syndrome,; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Since both pathologies (PCOS and NAFLD) involve disturbed carbohydrate economy, which revolve around insulin resistance, it is tempting to examine the specific "liver profile" of women with PCOD. Furthermore, it would be of great importance if lean women who suffer from PCOD would be revealed to shere cardiovascular risks with their more overweight peers.

Patients - women who will be diagnosed with PCOD following their initial referal to our fertility clinic. Controls - normal ovulatory women who approached our fertility clinic due to either unexplained or male factor infertility.

Workup - history for menstrual pattern; Clinical evaluation for features of hyperandrogenism; ultrasonographic documentation of ovarian morphology; follicular phase hormonal profile for validation of the diagnosis and for ruling out other pathologies which may cause anovulation.

Liver profiling - The following blood tests will be used for the biochemical profiling: fasting glucose and insulin, CRP, HDL-cholesterol, triglycerides, AST, ALT, GGT, LDH, alkaline phosphatase, total bilirubin, direct bilirubin, ferritin, HBA1C and micro albumin ratio.

FibroScan® will be used to measure liver stiffness.

ELIGIBILITY:
Workup - history for menstrual pattern; Clinical evaluation for features of hyperandrogenism; ultrasonographic documentation of ovarian morphology; follicular phase hormonal profile for validation of the diagnosis and for ruling out other pathologies which may cause anovulation.

Liver profiling - The following blood tests will be used for the biochemical profiling: fasting glucose and insulin, CRP, HDL-cholesterol, triglycerides, AST, ALT, GGT, LDH, alkaline phosphatase, total bilirubin, direct bilirubin, ferritin, HBA1C and micro albumin ratio.

FibroScan® will be used to measure liver stiffness, as previously described

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients - women who will be diagnosed with PCOD following their initial referal to our fertility clinic. Controls - normal ovulatory women who approached our fertility clinic due to either unexplained or male factor infertility.
Sampling Method: Non-Probability Sample
Dates: Start 2012-11

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Clinic, ZIv Medical Center, Safed, Israel